CLINICAL TRIAL: NCT03615794
Title: A Prospective Study of Pregnant and Postpartum Women With and Without Mood Disorders
Brief Title: A Study of Pregnant and Postpartum Women With and Without Mood Disorders
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00027369
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Postpartum Depression; Postpartum Psychosis
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will undergo a blood draw at every in-person visit. Whole blood for genetic/epigenetic studies, serum for hormonal and immunological makers, and blood for a Complete Blood Count (CBC) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with Mood Disorders: Pregnant women with a history or current diagnosis of Major Depressive Disorder or Bipolar Disorder
- Healthy controls: Pregnant women without a history or current diagnosis of a mood disorder.

SUMMARY:
This study is looking at genetic, biological, and environmental causes and how all three may work together to cause postpartum mood episodes. Participants will have psychiatric histories taken and will be monitored throughout pregnancy and during the postpartum period for the development of depressive or other mood episodes. Biological measures, including hormone levels, immunological measures, and growth factors will be collected. Environmental factors such as sleep deprivation and stress will also be measured. These factors will be considered in the setting of genetic and epigenetic data with the hope that investigators will ultimately be able to predict the onset of postpartum mood episodes in this vulnerable population.

DETAILED DESCRIPTION:
Postpartum Depression (PPD) is a serious syndrome which resembles a major depressive episode and occurs in 10-20% of all mothers in the year following delivery. In addition, 20 - 30 % of women with Bipolar Disorder will experience postpartum psychosis (mania) and at least 20 % will experience a postpartum depression with some estimates as high as 65%. The postpartum time therefore represents a natural experiment that, in the setting of prospective monitoring, will allow the measurement of biological, genetic, and environmental factors that may impact the development of mood episodes.

Data was previously collected in "A Prospective Study of Postpartum Mood Episodes in Women with Affective disorders." Investigators followed 93 women with a history of a mood disorder (Major Depressive Disorder, Bipolar I, Bipolar II or Bipolar Not Otherwise Specified) through pregnancy and up to three months postpartum. This was a very ill sample and around 75% of the participants met Diagnostic and Statistical Manual (DSM)-IV criteria for a Major Depressive Episode either during pregnancy, postpartum or both. Of those that were well during the 3rd trimester (N=38), 40% became depressed within 4 weeks of delivery, despite the fact that 80% were taking psychiatric medications. Of those that developed Postpartum Depression, 53% had a family history of Postpartum Depression compared to 12% of those that did not develop Postpartum Depression, thus demonstrating a potential genetic basis for Postpartum Depression. Using this sample, investigators were able to identify epigenetic biomarkers that were predictive of Postpartum Depressive episodes.

Investigators now seek to replicate and extend investigators' previous findings by identifying and following a second sample of women with mood disorders through pregnancy and into the postpartum time period and, in addition, collect a sample of pregnant women who do not have a history of mood disorder as a control sample. These women will have psychiatric histories taken and will be monitored throughout pregnancy and during the postpartum period for the development of depressive or other mood episodes. In addition to clinical data, biological measures such as hormone levels, immunological measures and growth factors will be taken. Environmental factors such as sleep deprivation and stress will also be measured. These factors will be considered in the setting of genetic and epigenetic data with the hope that investigators will ultimately be able to predict the onset of postpartum mood episodes in this vulnerable population. An understanding of the biological basis of postpartum episodes will ultimately shed light on the vulnerability to Major Depressive Disorder and Bipolar Disorder in general

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies
* With or without a history of a mood disorder (MDD, Bipolar I, Bipolar II or Bipolar NOS)

Exclusion Criteria:

* Current active suicidal ideation
* Medical or psychiatric instability
* Active substance abuse or dependence during the last 90 days
* Presence or development of significant pregnancy conditions that may have independent effects on outcomes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with or without a history of a mood disorder (Major Depression, Bipolar I, Bipolar II, or Bipolar NOS).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Major depressive episode | 4 weeks postpartum
  Development of a major depressive episode within the first 4 weeks postpartum

SECONDARY OUTCOMES:
Postpartum depression as assessed by Whole blood analysis | Pregnancy and up to 6 months postpartum
  Analyze whole blood to identify genetic and epigenetic risk factors for postpartum depression.
Postpartum depression risk as assessed by serum analysis | Pregnancy and up to 6 months postpartum
  Analyze serum samples to identify hormonal and immunological risk factors for postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Payne, MD, Principal Investigator — University of Virginia; Richard Lee, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - 550 North Broadway, Baltimore, Maryland
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akman I, Kuscu K, Ozdemir N, Yurdakul Z, Solakoglu M, Orhan L, Karabekiroglu A, Ozek E. Mothers' postpartum psychological adjustment and infantile colic. Arch Dis Child. 2006 May;91(5):417-9. doi: 10.1136/adc.2005.083790. Epub 2006 Feb 1. PMID 16452109
- [Background] Bernstein, D. and L. Fink, Manual for the childhood trauma questionnaire. The Psychological Corporation, New York, 1998
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Background] Bratfos O, Haug JO. Puerperal mental disorders in manic-depressive females. Acta Psychiatr Scand. 1966;42(3):285-94. doi: 10.1111/j.1600-0447.1966.tb01933.x. No abstract available. PMID 5959091
- [Background] Campbell SB, Cohn JF. Prevalence and correlates of postpartum depression in first-time mothers. J Abnorm Psychol. 1991 Nov;100(4):594-9. doi: 10.1037//0021-843x.100.4.594. PMID 1757673
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cohen LS, Nonacs RM, Bailey JW, Viguera AC, Reminick AM, Altshuler LL, Stowe ZN, Faraone SV. Relapse of depression during pregnancy following antidepressant discontinuation: a preliminary prospective study. Arch Womens Ment Health. 2004 Oct;7(4):217-21. doi: 10.1007/s00737-004-0059-3. Epub 2004 Aug 30. PMID 15338315
- [Background] Cohen LS, Altshuler LL, Harlow BL, Nonacs R, Newport DJ, Viguera AC, Suri R, Burt VK, Hendrick V, Reminick AM, Loughead A, Vitonis AF, Stowe ZN. Relapse of major depression during pregnancy in women who maintain or discontinue antidepressant treatment. JAMA. 2006 Feb 1;295(5):499-507. doi: 10.1001/jama.295.5.499. PMID 16449615
- [Background] Cox JL, Murray D, Chapman G. A controlled study of the onset, duration and prevalence of postnatal depression. Br J Psychiatry. 1993 Jul;163:27-31. doi: 10.1192/bjp.163.1.27. PMID 8353695
- [Background] Davidson J, Robertson E. A follow-up study of post partum illness, 1946-1978. Acta Psychiatr Scand. 1985 May;71(5):451-7. doi: 10.1111/j.1600-0447.1985.tb05057.x. PMID 4013805
- [Background] Dean C, Williams RJ, Brockington IF. Is puerperal psychosis the same as bipolar manic-depressive disorder? A family study. Psychol Med. 1989 Aug;19(3):637-47. doi: 10.1017/s0033291700024235. PMID 2798633
- [Background] Dietz PM, Williams SB, Callaghan WM, Bachman DJ, Whitlock EP, Hornbrook MC. Clinically identified maternal depression before, during, and after pregnancies ending in live births. Am J Psychiatry. 2007 Oct;164(10):1515-20. doi: 10.1176/appi.ajp.2007.06111893. PMID 17898342
- [Background] DiPietro JA, Costigan KA, Gurewitsch ED. Fetal response to induced maternal stress. Early Hum Dev. 2003 Nov;74(2):125-38. doi: 10.1016/j.earlhumdev.2003.07.001. PMID 14580752
- [Background] Field T. Prenatal depression effects on early development: a review. Infant Behav Dev. 2011 Feb;34(1):1-14. doi: 10.1016/j.infbeh.2010.09.008. PMID 20970195
- [Background] Flynn HA, Davis M, Marcus SM, Cunningham R, Blow FC. Rates of maternal depression in pediatric emergency department and relationship to child service utilization. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):316-22. doi: 10.1016/j.genhosppsych.2004.03.009. PMID 15234828
- [Background] Forty L, Jones L, Macgregor S, Caesar S, Cooper C, Hough A, Dean L, Dave S, Farmer A, McGuffin P, Brewster S, Craddock N, Jones I. Familiality of postpartum depression in unipolar disorder: results of a family study. Am J Psychiatry. 2006 Sep;163(9):1549-53. doi: 10.1176/ajp.2006.163.9.1549. PMID 16946179
- [Background] Frank E, Kupfer DJ, Jacob M, Blumenthal SJ, Jarrett DB. Pregnancy-related affective episodes among women with recurrent depression. Am J Psychiatry. 1987 Mar;144(3):288-93. doi: 10.1176/ajp.144.3.288. PMID 3826425
- [Background] Grace SL, Evindar A, Stewart DE. The effect of postpartum depression on child cognitive development and behavior: a review and critical analysis of the literature. Arch Womens Ment Health. 2003 Nov;6(4):263-74. doi: 10.1007/s00737-003-0024-6. PMID 14628179
- [Background] Guintivano J, Arad M, Gould TD, Payne JL, Kaminsky ZA. Antenatal prediction of postpartum depression with blood DNA methylation biomarkers. Mol Psychiatry. 2014 May;19(5):560-7. doi: 10.1038/mp.2013.62. Epub 2013 May 21. PMID 23689534
- [Background] 20) Guy W. Clinical global impression. ECDEU Assessment Manual for Psychopharmacology, Revised 1976, National Institute of Mental Health, Rockville, MD.
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Jones I, Middle F, McCandless F, Coyle N, Robertson E, Brockington I, Lendon C, Craddock N. Molecular genetic studies of bipolar disorder and puerperal psychosis at two polymorphisms in the estrogen receptor alpha gene (ESR 1). Am J Med Genet. 2000 Dec 4;96(6):850-3. doi: 10.1002/1096-8628(20001204)96:63.0.co;2-1. PMID 11121195
- [Background] Jones I, Craddock N. Familiality of the puerperal trigger in bipolar disorder: results of a family study. Am J Psychiatry. 2001 Jun;158(6):913-7. doi: 10.1176/appi.ajp.158.6.913. PMID 11384899
- [Background] Jones I, Hamshere M, Nangle JM, Bennett P, Green E, Heron J, Segurado R, Lambert D, Holmans P, Corvin A, Owen M, Jones L, Gill M, Craddock N. Bipolar affective puerperal psychosis: genome-wide significant evidence for linkage to chromosome 16. Am J Psychiatry. 2007 Jul;164(7):1099-104. doi: 10.1176/ajp.2007.164.7.1099. PMID 17606662
- [Background] Kendell RE, Chalmers JC, Platz C. Epidemiology of puerperal psychoses. Br J Psychiatry. 1987 May;150:662-73. doi: 10.1192/bjp.150.5.662. PMID 3651704
- [Background] Kimmel M, Hess E, Roy PS, Palmer JT, Meltzer-Brody S, Meuchel JM, Bost-Baxter E, Payne JL. Family history, not lack of medication use, is associated with the development of postpartum depression in a high-risk sample. Arch Womens Ment Health. 2015 Feb;18(1):113-21. doi: 10.1007/s00737-014-0432-9. Epub 2014 Jul 1. PMID 24980575
- [Background] Lee KA. Self-reported sleep disturbances in employed women. Sleep. 1992 Dec;15(6):493-8. doi: 10.1093/sleep/15.6.493. PMID 1475563
- [Background] Mahon PB, Payne JL, MacKinnon DF, Mondimore FM, Goes FS, Schweizer B, Jancic D; NIMH Genetics Initiative Bipolar Disorder Consortium; BiGS Consortium; Coryell WH, Holmans PA, Shi J, Knowles JA, Scheftner WA, Weissman MM, Levinson DF, DePaulo JR Jr, Zandi PP, Potash JB. Genome-wide linkage and follow-up association study of postpartum mood symptoms. Am J Psychiatry. 2009 Nov;166(11):1229-37. doi: 10.1176/appi.ajp.2009.09030417. Epub 2009 Sep 15. PMID 19755578
- [Background] Marcus SM. Depression during pregnancy: rates, risks and consequences--Motherisk Update 2008. Can J Clin Pharmacol. 2009 Winter;16(1):e15-22. Epub 2009 Jan 22. PMID 19164843
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Murphy-Eberenz K, Zandi PP, March D, Crowe RR, Scheftner WA, Alexander M, McInnis MG, Coryell W, Adams P, DePaulo JR Jr, Miller EB, Marta DH, Potash JB, Payne J, Levinson DF. Is perinatal depression familial? J Affect Disord. 2006 Jan;90(1):49-55. doi: 10.1016/j.jad.2005.10.006. Epub 2005 Dec 5. PMID 16337009
- [Background] Misri S, Eng AB, Abizadeh J, Blackwell E, Spidel A, Oberlander TF. Factors impacting decisions to decline or adhere to antidepressant medication in perinatal women with mood and anxiety disorders. Depress Anxiety. 2013 Nov;30(11):1129-36. doi: 10.1002/da.22137. Epub 2013 Jun 18. PMID 23780823
- [Background] O'Donnell KJ, Bugge Jensen A, Freeman L, Khalife N, O'Connor TG, Glover V. Maternal prenatal anxiety and downregulation of placental 11beta-HSD2. Psychoneuroendocrinology. 2012 Jun;37(6):818-26. doi: 10.1016/j.psyneuen.2011.09.014. Epub 2011 Oct 15. PMID 22001010
- [Background] 35) O'Hara MW, Varner, MW. (1986). Assessing stressful life events associated with childbearing: The Peripartum Events Scale. J of Repro and Inf Psych 4: 85-98.
- [Background] O'Hara MW. Postpartum depression: what we know. J Clin Psychol. 2009 Dec;65(12):1258-69. doi: 10.1002/jclp.20644. PMID 19827112
- [Background] Payne JL, Roy PS, Murphy-Eberenz K, Weismann MM, Swartz KL, McInnis MG, Nwulia E, Mondimore FM, MacKinnon DF, Miller EB, Nurnberger JI, Levinson DF, DePaulo JR Jr, Potash JB. Reproductive cycle-associated mood symptoms in women with major depression and bipolar disorder. J Affect Disord. 2007 Apr;99(1-3):221-9. doi: 10.1016/j.jad.2006.08.013. Epub 2006 Oct 2. PMID 17011632
- [Background] Payne JL, MacKinnon DF, Mondimore FM, McInnis MG, Schweizer B, Zamoiski RB, McMahon FJ, Nurnberger JI Jr, Rice JP, Scheftner W, Coryell W, Berrettini WH, Kelsoe JR, Byerley W, Gershon ES, DePaulo JR Jr, Potash JB. Familial aggregation of postpartum mood symptoms in bipolar disorder pedigrees. Bipolar Disord. 2008 Feb;10(1):38-44. doi: 10.1111/j.1399-5618.2008.00455.x. PMID 18199240
- [Background] Reich T, Winokur G. Postpartum psychoses in patients with manic depressive disease. J Nerv Ment Dis. 1970 Jul;151(1):60-8. doi: 10.1097/00005053-197007000-00008. No abstract available. PMID 5426650
- [Background] Shadigian E, Bauer ST. Pregnancy-associated death: a qualitative systematic review of homicide and suicide. Obstet Gynecol Surv. 2005 Mar;60(3):183-90. doi: 10.1097/01.ogx.0000155967.72418.6b. PMID 16570396
- [Background] Shivakumar G, Johnson NL, McIntire DD, Leveno K. Progression of major depression during pregnancy and postpartum: a preliminary study. J Matern Fetal Neonatal Med. 2014 Apr;27(6):571-6. doi: 10.3109/14767058.2013.825599. Epub 2013 Aug 19. PMID 23865695
- [Background] Sichel DA, Cohen LS, Robertson LM, Ruttenberg A, Rosenbaum JF. Prophylactic estrogen in recurrent postpartum affective disorder. Biol Psychiatry. 1995 Dec 15;38(12):814-8. doi: 10.1016/0006-3223(95)00063-1. PMID 8750040
- [Background] Sit DK, Perel JM, Helsel JC, Wisner KL. Changes in antidepressant metabolism and dosing across pregnancy and early postpartum. J Clin Psychiatry. 2008 Apr;69(4):652-8. doi: 10.4088/jcp.v69n0419. PMID 18426260
- [Background] Somerville S, Dedman K, Hagan R, Oxnam E, Wettinger M, Byrne S, Coo S, Doherty D, Page AC. The Perinatal Anxiety Screening Scale: development and preliminary validation. Arch Womens Ment Health. 2014 Oct;17(5):443-54. doi: 10.1007/s00737-014-0425-8. Epub 2014 Apr 4. PMID 24699796
- [Background] Spinelli MG. Maternal infanticide associated with mental illness: prevention and the promise of saved lives. Am J Psychiatry. 2004 Sep;161(9):1548-57. doi: 10.1176/appi.ajp.161.9.1548. PMID 15337641
- [Background] Viguera AC, Tondo L, Koukopoulos AE, Reginaldi D, Lepri B, Baldessarini RJ. Episodes of mood disorders in 2,252 pregnancies and postpartum periods. Am J Psychiatry. 2011 Nov;168(11):1179-85. doi: 10.1176/appi.ajp.2011.11010148. Epub 2011 Jul 28. PMID 21799064
- [Background] Wisner KL, Wheeler SB. Prevention of recurrent postpartum major depression. Hosp Community Psychiatry. 1994 Dec;45(12):1191-6. doi: 10.1176/ps.45.12.1191. PMID 7868100
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH, Findling RL, Rapport D. Prevention of recurrent postpartum depression: a randomized clinical trial. J Clin Psychiatry. 2001 Feb;62(2):82-6. doi: 10.4088/jcp.v62n0202. PMID 11247106
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH, Piontek CM, Findling RL. Prevention of postpartum depression: a pilot randomized clinical trial. Am J Psychiatry. 2004 Jul;161(7):1290-2. doi: 10.1176/appi.ajp.161.7.1290. PMID 15229064
- [Background] Yonkers KA, Ramin SM, Rush AJ, Navarrete CA, Carmody T, March D, Heartwell SF, Leveno KJ. Onset and persistence of postpartum depression in an inner-city maternal health clinic system. Am J Psychiatry. 2001 Nov;158(11):1856-63. doi: 10.1176/appi.ajp.158.11.1856. PMID 11691692
- [Background] Yonkers KA, Gotman N, Smith MV, Forray A, Belanger K, Brunetto WL, Lin H, Burkman RT, Zelop CM, Lockwood CJ. Does antidepressant use attenuate the risk of a major depressive episode in pregnancy? Epidemiology. 2011 Nov;22(6):848-54. doi: 10.1097/EDE.0b013e3182306847. PMID 21900825
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692